CLINICAL TRIAL: NCT00640081
Title: A Two-arm Phase II Randomised Trial of Intermittent Chemotherapy Plus Continuous Cetuximab and of Intermittent Chemotherapy Plus Intermittent Cetuximab in First Line Treatment of Patients With K-ras-normal (Wild-type) Metastatic Colorectal Cancer
Brief Title: Combination Chemotherapy and Cetuximab as First-Line Therapy in Treating Patients With Advanced and/or Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cheryl Pugh (Other Government)
Responsible Party: Sponsor-Investigator, Cheryl Pugh, Clinical Project manager for COINB for Sponsor, Medical Research Council
Organization: Medical Research Council (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000589635; MRC-CTU-COIN-B/CR11; EUDRACT:2006-003049-17; ISRCTN38375681; EU-20828; MERCK-MRC-CTU-COIN-B/CR11
Record Dates: First submitted 2008-03-19; First posted 2008-03-20 (Estimated); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the colon; stage IV colon cancer; adenocarcinoma of the rectum; stage IV rectal cancer; stage III colon cancer; stage III rectal cancer; recurrent colon cancer; recurrent rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Capecitabine; Fluorouracil; Leucovorin; Oxaliplatin; Immunohistochemistry

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- D (Active Comparator): Intermittent chemotherapy plus intermittent cetuximab treatment comprising 12 weeks of chemotherapy plus cetuximab followed by a period off all therapy, with reintroduction of the same chemotherapy and cetuximab regimen for a further 12 weeks after initial progression off treatment
  Interventions: Biological: cetuximab; Drug: capecitabine; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis
- E (Experimental): Intermittent chemotherapy plus continuous cetuximab treatment comprising 12 weeks of chemotherapy plus cetuximab followed by a period of withdrawal of the chemotherapy, but continued weekly cetuximab monotherapy (maintenance cetuximab), with reintroduction of the same chemotherapy regimen to the cetuximab for a further 12 weeks after initial progression off chemotherapy treatment
  Interventions: Biological: cetuximab; Drug: capecitabine; Drug: fluorouracil; Drug: leucovorin calcium; Drug: oxaliplatin; Other: immunohistochemistry staining method; Other: laboratory biomarker analysis

INTERVENTIONS:
Biological: cetuximab
Drug: capecitabine
Drug: fluorouracil
Drug: leucovorin calcium
Drug: oxaliplatin
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. It is not yet known whether giving combination chemotherapy together with intermittent cetuximab is more effective than combination chemotherapy given together with continuous cetuximab in treating colorectal cancer.

PURPOSE: This randomized phase II trial is studying giving combination chemotherapy together with intermittent cetuximab to see how well it works compared to combination chemotherapy given together with continuous cetuximab as first-line therapy in treating patients with advanced or metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To compare the activity, in terms of failure-free survival, of patients with K-ras-normal (wild type) advanced and/or metastatic colorectal cancer treated with intermittent combination chemotherapy comprising oxaliplatin, leucovorin calcium, and fluorouracil (OxMdG) or oxaliplatin and capecitabine (XELOX) and intermittent vs continuous cetuximab as first-line therapy.
* To compare the safety and feasibility of these regimens in these patients.

Secondary

* To compare the safety of cetuximab reintroduction, in terms of frequency of grade 3-4 allergic reactions in these patients.
* To compare improvement in disease control (i.e., complete response plus partial response plus stable disease) at 24 weeks in patients treated with these regimens.
* To compare overall and progression-free survival of patients treated with these regimens.
* To compare response rates at 12, 24, and 36 weeks in patients treated with these regimens.
* To compare toxicity of these regimens in these patients.

OUTLINE: This is a multicenter study. Patients are randomised to 1 of 2 treatment arms.

* Arm I (intermittent chemotherapy and intermittent cetuximab): Patients receive 1 of the following combination chemotherapy and cetuximab regimens:

  * OxMdG: Patients receive oxaliplatin IV over 2 hours and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1 and 2. Patients also receive cetuximab IV over 1-2 hours on days 1 and 8. Treatment repeats every 14 days for up to 6 courses (12 weeks) in the absence of disease progression or unacceptable toxicity.
  * XELOX (for patients with line-related problems): Patients receive oxaliplatin IV over 2 hours on day 1 and oral capecitabine twice daily on days 1-15 (28 doses). Patients also receive cetuximab IV over 1-2 hours on days 1, 8, and 15. Treatment repeats every 21 days for up to 4 courses (12 weeks) in the absence of disease progression or unacceptable toxicity.

After completion of 12 weeks of study therapy, patients with disease progression are removed from study. Patients with stable or responding disease stop treatment with OxMdG or XELOX and cetuximab and undergo clinical evaluation at least every 6 weeks until disease progression or clinical deterioration. Upon evidence of disease progression or clinical deterioration, patients restart treatment with OxMdG or XELOX and cetuximab as before and continue to alternate 12 weeks of treatment with treatment breaks in the absence of disease progression or unacceptable toxicity. Patients with disease progression during study therapy stop treatment and proceed to second-line therapy or best supportive care.

* Arm II (intermittent chemotherapy and continuous cetuximab): Patients receive OxMdG or XELOX and cetuximab for 12 weeks as in arm I. Patients with disease progression after 12 weeks of study therapy are removed from study. Patients with stable or responding disease* after 12 weeks of study therapy stop treatment with OxMdG or XELOX and continue treatment with cetuximab weekly as monotherapy in the absence of disease progression or unacceptable toxicity. Patients undergo clinical evaluation as in arm I. Upon progression, patients restart treatment with OxMdG or XELOX and continue cetuximab, as before, alternating 12 weeks of combined OxMdG or XELOX and cetuximab therapy with cetuximab monotherapy. Patients with disease progression during study therapy stop treatment and proceed to second-line therapy as in arm I.

Previously collected tumor tissue samples are obtained at baseline and analyzed by IHC for EGFR status of tumor.

After completion of study treatment, patients are followed every 12 weeks.

Peer Reviewed and Funded or Endorsed by Cancer Research UK.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of colorectal adenocarcinoma, defined by 1 of the following:

  * Prior or current histologically confirmed primary adenocarcinoma of colon or rectum with clinical or radiological evidence of advanced and/or metastatic disease
  * Histologically and cytologically confirmed metastatic adenocarcinoma with clinical and/or radiological evidence of colorectal primary tumor
* Unidimensionally measurable disease by RECIST criteria
* Inoperable metastatic or locoregional disease

  * Potentially resectable liver metastases allowed provided the following criteria are met:

    * Fewer than 4 unilobar liver metastases, each < 4 cm in size and without major vascular involvement
    * No combination chemotherapy allowed prior to the planned resection of operable liver metastases
* No confirmed K-ras mutation of tumor after screening
* No brain metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-2
* Must be considered fit to undergo combination chemotherapy
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Serum bilirubin ≤ 1.25 times upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 times ULN
* AST or ALT ≤ 2.5 times ULN
* Creatinine clearance ≥ 50mL/min OR glomerular filtration rate ≥ 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No severe uncontrolled concurrent medical illness (including poorly controlled angina or myocardial infarction within the past 12 weeks) likely to interfere with protocol treatments
* No psychiatric or neurological condition that would preclude study compliance with oral medication or giving informed consent
* No partial or complete bowel obstruction
* No preexisting neuropathy > grade 1
* No prior or current malignant disease which, in the judgement of the treating investigator, is likely to interfere with COIN-B treatment or assessment of response
* No patients with known hypersensitivity reactions to any of the components of the study treatments
* No proven dihydropyrimidine dehydrogenase deficiency (DPD) or personal or family history of DPD

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior systemic palliative chemotherapy for metastatic disease
* No prior oxaliplatin
* More than 1 month since prior adjuvant chemotherapy comprising fluorouracil (with or without leucovorin calcium), capecitabine, or irinotecan hydrochloride
* More than 1 month since prior chemoradiotherapy comprising fluorouracil (with or without leucovorin calcium) or capecitabine for rectal cancer
* No ongoing requirement for contraindicated concurrent medication
* No concurrent enrollment in any type of study other than observational studies

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2007-07; Primary Completion 2010-06 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Failure-free survival at 10 months | 10 months

SECONDARY OUTCOMES:
Safety of cetuximab reintroduction, in terms of risk of grade 3-4 allergic reactions | 12, 24 and 36 weeks
Proportion of patients achieving disease control (complete response plus partial response plus stable disease) at 24 weeks | 24 weeks
Overall survival | at 12, 24 and 36 weeks
Progression-free survival | at 12, 24 and 36 weeks
Response rates | at 12, 24 and 36 weeks
Toxicity of each treatment regimen by NCI CTCAE v3.0 | at 12, 24 and 36 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harpreet S. Wasan, Principal Investigator — Hammersmith Hospitals NHS Trust
Locations (25):
- Bank of Cyprus Oncology Centre, Nicosia, Cyprus
- United Kingdom (24):
  - Bradford Royal Infirmary, Bradford, England
  - Gloucestershire Oncology Centre at Cheltenham General Hospital, Cheltenham, England
  - Essex County Hospital, Colchester, England
  - Dorset County Hospital, Dorchester, England
  - St. Luke's Cancer Centre at Royal Surrey County Hospital, Guildford, England
  - Hammersmith Hospital, London, England
  - St. Mary's Hospital, London, England
  - Churchill Hospital, Oxford, England
  - Peterborough Hospitals Trust, Peterborough, England
  - University Hospital of North Staffordshire, Stoke-on-Trent, England
  - Singleton Hospital, Swansea, Wales
  - Royal United Hospital, Bath
  - Royal Bournemouth Hospital, Bournemouth
  - Addenbrookes Hospital, Cambridge
  - Darent Valley Hospital, Dartford
  - Hereford County Hospital, Hereford
  - Charing Cross Hospital, London
  - Guys and St Thomas' hospitals, London
  - Dorset Cancer Centre, Poole Hospital, Poole
  - Weston Park, Sheffield
  - Southport and Ormskirk, Southport
  - St Helens and Whiston hospitals, St Helens
  - Warrington and Halton Hospitals, Warrington
  - Worcestershire Royal Hospital, Worcester

IPD SHARING:
Plan to Share IPD: Yes
Publication
URL: http://www.thelancet.com/journals/lanonc/article/PIIS1470-2045(14)70106-8/abstract

REFERENCES:
- See also: Trial Summary on Sponsor's Website with trial citations — http://www.ctu.mrc.ac.uk/our_research/research_areas/cancer/studies/coin_b/